CLINICAL TRIAL: NCT06382831
Title: Comparing Opioid Free Versus Opioid Balanced Anesthesia in Ophthalmic Surgery: a Single Centre Randomized Controlled Trial
Brief Title: Opioid Free Versus Opioid Balanced Anesthesia in Ophthalmic Surgery
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IndonesiaU240201
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia and Analgesia; Anesthesia, Endotracheal
Keywords: Opioid free anesthesia; Ocular surgery; Ophthalmology surgery; Dexmedetomidine; Post operative nausea and vomiting
MeSH Terms: conditions — Agnosia; Vomiting | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Fentanyl
- Opioid free anesthesia (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Opioid free anesthesia
  Arms: Opioid free anesthesia
Drug: Fentanyl — Control given Opioid balanced anesthesia
  Arms: Control

SUMMARY:
Anesthesia without the use of opioid (Opioid free anesthesia) is an alternative to conventional opioid balanced anesthesia, with less post operative nausea and vomiting, and comparable analgesia. This study aim to compare the effect of opioid free versus opioid balanced anesthesia in ophthalmology surgery

ELIGIBILITY:
Inclusion Criteria:

* Physical status of ASA 1-2
* Undergo elective ophthalmology surgery under general anesthesia with laryngeal mask insertion
* BMI 17.5-34.9

Exclusion Criteria:

* Allergy to study drugs
* Baseline heart rate < 70 beat per minute or systolic blood pressure < 100 mmHg
* Will undergo regional block
* Operation lasting for > 4 hours or < 90 minutes
* Consumes opioid routinely prior to operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 hours
  Incidence of PONV
Pain score | 24 hours
  Pain score assessed with numerical rating scale (0-10) where higher value corresponds to more pain experienced by the patient
Time to laryngeal mask exertion | Intraoperative
  Measured from the last surgical knot to LMA exertion
Adverse effect | 24 hours
  Severe changes in hemodynamics, including severe bradycardia, tachycardia, hypotension, hypertension, desaturation

IPD SHARING:
Plan to Share IPD: No
Participants' data is kept under strict regulation by the study investigator and will not be shared without participants' consent